CLINICAL TRIAL: NCT01790178
Title: Outcomes of Ultrasound-guided Versus Blind Core Muscle Biopsy
Brief Title: Ultrasound in Muscle Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Pro00041999
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Myopathy; Myositis; Muscular Dystrophy
MeSH Terms: conditions — Muscular Diseases; Myositis; Muscular Dystrophies | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound Guided Biopsy (Experimental): Ultrasound guided biopsy will be used in all patients.
  Interventions: Procedure: Ultrasound
- Non-Ultrasound Guided Group (No Intervention): The control group will have non-ultrasound guided biopsies performed, which is the current standard of care.

INTERVENTIONS:
Procedure: Ultrasound — The ultrasound guided group will have an ultrasound to identify the optimal site for biopsy and guide the procedure for safety purposes.
  Arms: Ultrasound Guided Biopsy

SUMMARY:
The objective of the proposed study is to evaluate the clinical utility of muscle ultrasonography for improving the diagnostic yield and safety of core muscle biopsy. Our facility currently uses core (needle) biopsy to obtain muscle samples in patients 18 years old or older. Currently, there is no imaging tool used to guide the actual biopsy. As muscle biopsy is an invasive and potentially painful procedure, improving the diagnostic yield of this test is important.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive subjects scheduled for a biopsy at our EMG laboratory will be asked if they would like to participate until a total of 40 participants are obtained.

Exclusion Criteria:

* Age under 18 years.
* Inability to provide consent for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D. Hobson-Webb, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound Guided Biopsy | Non-Ultrasound Guided Group
Started | 16 | 24
Completed | 16 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound Guided Biopsy | Non-Ultrasound Guided Group | Total
Number analyzed (Participants) | 16 | 24 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 21 | 27
  >=65 years | 10 | 3 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1875 (19.8) | 55.375 (12.8) | 55.7 (15.7)
Gender [Count of Participants; unit: Participants]
  Female | 9 | 17 | 26
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 16 | 24 | 40

OUTCOME MEASURES:

1. Primary Outcome: Amount of Tissue Obtained
Description: This data will be analyzed to determine if ultrasound guidance improves muscle yield (as measured by pathology determined volume and mass).
Time Frame: At time of biopsy
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Ultrasound Guided Biopsy | Non-Ultrasound Guided Group
Number analyzed (Participants) | 16 | 24
grams | 0.29 (0.23) | 0.28 (0.21)

2. Primary Outcome: Number of Patients Receiving Diagnosis From Muscle Biopsy
Description: The rate of achieving a specific final diagnosis in ultrasound guided muscle biopsies vs. unguided biopsies will be examined.
Time Frame: At time of biopsy
Measure: Number; unit: participants
Arm/Group | Ultrasound Guided Biopsy | Non-Ultrasound Guided Group
Number analyzed (Participants) | 16 | 24
participants | 7 | 12

3. Secondary Outcome: Number of Participants With Adverse Events Related to Muscle Biopsy
Description: Data will be examined to determine if ultrasound guidance reduces the rate of adverse events in muscle biopsies.
Time Frame: Patient involvement limited to the time of biopsy; Records analyzed up to 10 months after biopsy
Measure: Number; unit: participants
Arm/Group | Ultrasound Guided Biopsy | Non-Ultrasound Guided Group
Number analyzed (Participants) | 16 | 24
participants | 0 | 0

4. Secondary Outcome: Number of Times Biopsy Needle Was Inserted to Obtain Biopsy Tissue
Description: For "core" or "needle" biopsies, the physician passes the needle into the muscle until they feel that adequate tissue samples have been obtained. This outcome measure is the number of passes required in each study arm.
Time Frame: At time of biopsy
Measure: Mean (Standard Deviation); unit: needle passes
Arm/Group | Ultrasound Guided Biopsy | Non-Ultrasound Guided Group
Number analyzed (Participants) | 16 | 24
needle passes | 2.57 (0.756) | 2.5 (0.761)

5. Secondary Outcome: Number of Participants With Inadequate Biopsy Samples
Description: The presence of an inadequate sample was determined by the blinded pathologist reading the muscle biopsies. This reflects the sample having enough preserved muscle tissue for histologic analysis. It is separate from the number of participants receiving a diagnosis. A sample may be adequate, but non-diagnostic. Only one biopsy was performed in each patients, so the number of biopsies is the same as the number of participants.
Time Frame: At time of pathology review
Measure: Number; unit: Inadequate Biopsy Samples
Arm/Group | Ultrasound Guided Biopsy | Non-Ultrasound Guided Group
Number analyzed (Participants) | 16 | 24
Inadequate Biopsy Samples | 1 | 2

ADVERSE EVENTS:
Time Frame: Time of consent to Six months
Arm/Group | Ultrasound Guided Biopsy | Non-Ultrasound Guided Group
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/24
Other Adverse Events (participants affected / at risk) | 0/16 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No